CLINICAL TRIAL: NCT02328300
Title: FLT PET/MR for Evaluation of Pseudoprogression in Patients With Brain Lesions
Status: Withdrawn | Type: Observational
Why Stopped: FLT production not available
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1327
Record Dates: First submitted 2014-08-29; First posted 2014-12-31 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Brain Lesions; Brain Metastasis; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FLT PET/MR: All participants will have known brain lesion in the central nervous system (CNS) scheduled to have surgical biopsy of the lesion, identified by the UNC Brain Tumor Board and will have the clinical question of radiation necrosis vs. recurrence.
  All participants will receive a FLT PET/MR scan.
  Interventions: Drug: FLT PET/MR

INTERVENTIONS:
Drug: FLT PET/MR — Each participant will be injected with FLT, a common PET radiotracer for brain tumors and lesions, and then will complete one (1) PET/MR scan.
  Other Names: FLT PET/MRI

SUMMARY:
This is a single arm, single center study of 15 patients with brain lesions being treated at UNC Hospitals. Subjects will undergo one (1) FLT-PET-MRI scan before their scheduled surgical biopsy of their brain lesion(s).

DETAILED DESCRIPTION:
Identifying imaging biomarkers of metastatic brain tumor treatment response could allow early modification of treatment by determination of tumor progression vs. treatment related effects (pseudo-progression, radiation necrosis). Earlier treatment response assessment could reduce cost, improve clinical trial efficiency and allow better assessment of prognosis. The development of PET/MRI offers the possibility of combining the functional imaging of PET with the exquisite soft tissue contrast and physiologic imaging capabilities of MRI. Combining FLT-PET imaging with MRI may allow better evaluation of new and unclear lesions in brain metastatic disease. The goal of this study is to explore FLT-PET imaging combined with dynamic MR imaging techniques for the identification of tumor response markers in metastatic brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Known brain lesion in central nervous system (CNS) scheduled to have surgical biopsy of the lesion, identified by the UNC Brain Tumor Board as having clinical question of radiation necrosis vs. recurrence
* At least one measurable lesion greater than 1 cm in diameter
* ≥ 18 years of age
* Study-specific informed consent reviewed and signed

Exclusion Criteria:

* Pregnant, nursing, or planning to become pregnant within 30 days of anticipated PET-MRI scan
* Condition that makes MRI unsafe (e.g., cardiac pacemaker, epicardial pacemaker leads, cochlear implants, metal aneurysm clips, metal halo devices)
* Inability to tolerate MRI (e.g., unable to lie flat for > 1 hour, severe claustrophobia)
* Allergy to MRI contrast agent (Magnevist, Multihance, Ablavar, Dotarem, Eovist, Gadavist)
* Known allergy to fluorothymidine
* Study participation would cause significant delay (> 2 weeks) in scheduled standard of care therapy
* Creatinine clearance < 60 ml/min, as estimated by the Cockcroft-Gault formula
* Body Mass Index (BMI) > 35
* Poorly controlled diabetes mellitus (fasting blood glucose > 200 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UNC Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of FLT-PET-MRI in distinguishing between recurrence and radiation necrosis, with surgical biopsy as gold standard | 1 week post-surgical biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Lee, MD/PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States